CLINICAL TRIAL: NCT03201718
Title: Post-marketing Surveillance Study of Viekira/ Exviera Tablets for Korean Hepatitis C Patients According to the Standard for "Re-examination of New Drugs"
Brief Title: A Study of Viekira/Exviera for Korean Hepatitis C Patients According to the Standard for Re-examination of New Drugs
Acronym: HCV PMS
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P16-666
Record Dates: First submitted 2017-06-27; First posted 2017-06-28 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Hepatitis C Virus (HCV)
Keywords: Hepatitis C; Paritaprevir; Ritonavir; Ombitasvir; Dasabuvir
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hepatitis C: Participants with Hepatitis C receiving Viekira/Exviera (paritaprevir/ritonavir/ombitasvir and dasabuvir) for 12 or 24 weeks.

SUMMARY:
Post-marketing surveillance study to evaluate the real world safety and effectiveness of Viekira/ Exviera (paritaprevir/ritonavir/ombitasvir and dasabuvir) administered under a normal, routine treatment practice by Korean patients with Hepatitis C.

ELIGIBILITY:
Inclusion Criteria:

* Participants with type C hepatitis
* Participants prescribed Viekira/Exviera in accordance with approved local label

Exclusion Criteria:

* None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type C Hepatitis patients who had been prescribed Viekira/Exviera (paritaprevir/ritonavir/ombitasvir and dasabuvir) in accordance with approved local label.
Sampling Method: Probability Sample
Enrollment: 505 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Sustained Virological Response 12 Weeks Post-treatment (SVR12) | 12 weeks after the last dose of study drug
  the lower limit of quantitation (LLOQ) SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 12 weeks after the last dose of study drug.

SECONDARY OUTCOMES:
Percentage of Participants With On-treatment Virologic Failure | Up to 24 weeks
  On-treatment virologic failure was defined as confirmed HCV RNA ≥ LLOQ after HCV RNA < LLOQ during treatment; confirmed increase of > 1 log(subscript)10(subscript) IU/mL above the lowest value post-baseline in HCV RNA during treatment; or HCV RNA ≥ LLOQ at end of treatment with at least 6 weeks of treatment.
Percentage of Participants With Post-treatment Relapse | From the end of treatment through 12 weeks after the last dose of study drug
  Post-treatment relapse defined as confirmed HCV RNA ≥ LLOQ between end of treatment and 12 weeks after the last dose of study drugs among participants who complete treatment and with HCV RNA levels < LLOQ at the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (59):
- South Korea (59):
  - Dong-A University Hospital /ID# 167362, Busan, Busan Gwang Yeogsi
  - Pusan National University Hosp /ID# 167363, Busan, Busan Gwang Yeogsi
  - Kyungpook National Univ Hosp /ID# 168731, Daegu, Daegu Gwang Yeogsi
  - Yeungnam University Med Ctr /ID# 167425, Daegu, Daegu Gwang Yeogsi
  - Chungnam National University Hospital /ID# 167724, Junggu, Daejeon Gwang Yeogsi
  - National health insurance cooperation ilsan hospital /ID# 201806, Goyang, Gyeonggido
  - Soon Chun Hyang University Hospital Bucheon /ID# 201803, Habun, Gyeonggido
  - Seoul National Univ Bundang ho /ID# 167394, Seongnam, Gyeonggido
  - St. Vincent's Hospital /ID# 201660, Suwon, Gyeonggido
  - Ajou University Hospital /ID# 167729, Suwon, Gyeonggido
  - Inje University Busan Paik Hospital /ID# 167392, Pusan, Gyeongsangbuk-do
  - Changwon Fatima Hospital /ID# 201664, Changwon, Gyeongsangnam-do
  - Inha University Hospital /ID# 201802, Junggu, Incheon Gwang Yeogsi
  - Chonnam National University Hospital /ID# 167423, Gwangju, Jeonranamdo
  - Kwangju Christian Hospital /ID# 210823, Gwangju, Jeonranamdo
  - Kyungpook National University Chilgok Hospital /ID# 201804, Daegu, Seoul Teugbyeolsi
  - SMG-SNU Boramae Medical Center /ID# 201805, Dongjak-gu, Seoul Teugbyeolsi
  - Kangbuk Samsung Hospital /ID# 168792, Jongno-Gu, Seoul Teugbyeolsi
  - Severance Hospital /ID# 167361, Seoul, Seoul Teugbyeolsi
  - Konkuk University Medical Ctr /ID# 167723, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 167722, Seoul, Seoul Teugbyeolsi
  - Korea Universtiy Guro Hospital /ID# 167388, Seoul, Seoul Teugbyeolsi
  - Bucheon St. Mary's hospital /ID# 170782, Bucheon-si
  - Dongnam Institute of Radiologi /ID# 167721, Busan
  - Good Samsun Hospital /ID# 167365, Busan
  - Haeundae Paik Hospital /ID# 170767, Busan
  - Maryknoll Medical Center /ID# 167418, Busan
  - Kosin University Gospel Hosp /ID# 168797, Busan
  - Samsung Changwon Hospital /ID# 167732, Changwon
  - Dankook University Hospital /ID# 167730, Cheonan
  - Chuncheon Sacred Heart Hosp /ID# 167419, Chuncheon
  - Kim Jun Hwan Sok Internal Medi /ID# 168794, Daegu
  - Keimyung Univ Dongsan medical /ID# 168793, Daegu
  - Daegu Catholic University Med /ID# 167714, Daegu
  - Daegu Catholic University Med /ID# 168729, Daegu
  - The Catholic Univ. of Korea /ID# 167733, Daejeon
  - Dongguk University Ilsan Hosp /ID# 168795, Goyang
  - Myongji Hospital /ID# 170784, Goyang
  - CHA Gumi Medical Center /ID# 170783, Gumi
  - Korea University Ansan Hosp /ID# 201661, Gyeonggi-do
  - Dongtan Sacred Heart Hospital /ID# 170759, Hwaseong
  - The Catholic University of Korea Incheon St.Mary's Hospital /ID# 170769, Incheon
  - Presbyterian Medical Center /ID# 167424, Jeonju
  - CHA Bundang Medical Center /ID# 170757, Seongnam
  - Bundang Jesaeng hospital /ID# 167725, Seongnam
  - Korea University Anam Hospital /ID# 167731, Seoul
  - Seoul National University Hospital /ID# 167364, Seoul
  - Seoul National University Hospital /ID# 167389, Seoul
  - SoonChunHyang University Seoul /ID# 167711, Seoul
  - Asan Medical Center /ID# 167390, Seoul
  - Chung-Ang University Hostipal /ID# 167420, Seoul
  - Inje University Seoul Paik Hos /ID# 167426, Seoul
  - Inje University Sanggye Paik H /ID# 167427, Seoul
  - St. Carollo General Hospital /ID# 167712, Suncheon
  - Uijeongbu St. Mary's Hospital /ID# 168730, Uijeongbu-si
  - Ulsan University Hospital /ID# 168796, Ulsan
  - Wonju Severance Christian Hosp /ID# 167713, Wŏnju
  - Pusan National University Yang /ID# 167710, Yangsan
  - Yeosoo Hankook Hospital /ID# 168728, Yeosu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/clinical-trials/ombitasvir_dasabuvir_P16-666.pdf